CLINICAL TRIAL: NCT06199908
Title: First-in-Human, Phase 1 Study of AMT-562 in Patients With Advanced Solid Tumors
Brief Title: AMT-562 in Patients With Selected Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Multitude Therapeutics (Australia) Pty Ltd (Industry)
Responsible Party: Sponsor
Organization: Multitude Therapeutics Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMT-562-01
Record Dates: First submitted 2023-12-21; First posted 2024-01-10 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2023-12

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): AMT-562 Dose Escalation
  Interventions: Drug: AMT-562

INTERVENTIONS:
Drug: AMT-562 — Administered AMT-562 for injection intravenously

SUMMARY:
This is a first-in-human, non-randomized, open-label, multicenter Phase 1 study of AMT-562 in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients must be willing and able to understand and sign the ICF, and to adhere to the study visit schedule and other protocol requirements.
* 2. Age ≥18 years (at the time consent is obtained).
* 3. Patients with histologically confirmed unresectable advanced solid tumor.
* 4. Patients who have undergone at least one systemic therapy and have radiologically or clinically determined progressive disease (PD) during or after most recent line of therapy, and for whom no further standard therapy is available, or who are intolerable to standard therapy.
* 5. Patients must have at least one measurable lesion as per RECIST version 1.1.
* 6. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* 7. Life expectancy ≥ 3 months.
* 8. Patients must have adequate organ function
* 9. Women of child bearing potential (WCBP), defined as a sexually mature woman who has not undergone surgical sterilization or who has not been naturally postmenopausal for at least 12 consecutive months (i.e., who has had menses any time in the preceding 12 consecutive months) must agree to use two effective contraceptive methods while on study treatment and for at least twelve weeks after the last dose of the IMP.
* 10. WCBP must have a negative serum pregnancy test within 7 days prior to first dose of the IMP.
* 11. Male patients must agree to use a latex condom, even if they had a successful vasectomy, while on study treatment and for at least twelve weeks after the last dose of the IMP.
* 12. Male patients must agree not to donate sperm, and female patients must agree not to donate eggs, while on study treatment and for at least 12 weeks after the last dose of the IMP.
* 13. Availability of tumor tissue sample (either an archival specimen or a fresh biopsy material) at screening.

Exclusion Criteria:

* 1. Central nervous system (CNS) metastasis.
* 2. Active or chronic skin disorder requiring systemic therapy.
* 3. History of Steven's Johnson's syndrome or toxic epidermal necrolysis syndrome.
* 4. Persistent toxicities from previous systemic anti-neoplastic treatments of Grade >1.
* 5. Systemic anti-neoplastic therapy within five half-lives or 21 days, whichever is shorter, prior to first dose of the IMP.
* 6. Radiotherapy to lung field at a total radiation dose of ≥ 20 Gy within 6 months, wide-field radiotherapy within 28 days.
* 7. Major surgery within 28 days prior to first dose of the IMP, or no recovery from side effects of such intervention.
* 8. Significant cardiac disease.
* 9. Has a history of (non-infectious) interstitial lung disease (ILD)/pneumonitis t.
* 10. History of thromboembolic or cerebrovascular events, including transient ischemic attacks, cerebrovascular accidents, deep vein thrombosis, or pulmonary emboli within six months prior to first dose of the IMP.
* 11. Acute and/or clinically significant bacterial, fungal or viral infection including hepatitis B (HBV), hepatitis C (HCV), known human immunodeficiency virus (HIV).
* 12. Administration of a live vaccine within 28 days prior to the administration of the first dose of the IMP.
* 13. Patients requiring concurrent treatment of strong inhibitors or inducers of cytochrome P450 3A or 1A2 enzyme (CYP3A or CYP1A2) within 2 weeks prior to the first dose and during the study treatment.
* 14. Known or suspected severe allergy/hypersensitivity (resulting in treatment discontinuation) to monoclonal antibodies.
* 15. Known or suspected intolerance to the components of the IMP.
* 16. Concurrent participation in another investigational therapeutic clinical trial.
* 17. Patients with known active alcohol or drug abuse.
* 18. Pregnant or breast-feeding females.
* 19. Mental or medical conditions that prevent the patient from giving informed consent or complying with the trial or other severe acute or chronic medical or psychiatric conditions or laboratory abnormality that may increase the risk associated with the study participation or the IMP administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for enrolment in this study.
* 20. Prior history of malignancy other than inclusion diagnosis within five years prior to first dose of the IMP.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-05-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
DLTs | up to 24 month
  Incidence of dose limiting toxicities
AEs | up to 24 month
  Type, incidence and severity of Adverse Events
SAEs | up to 24 month
  Type, incidence and severity Serious Adverse Events (SAEs)

SECONDARY OUTCOMES:
Cmax | up to 24 month
  Maximum concentration (Cmax)
Tmax | up to 24 month
  time to peak drug concentration
AUC | up to 24 month
  Area Under the Curve
t1/2 | up to 24 month
  terminal half-life of the ADC, total antibody and free payload
ADAs | up to 24 month
  Specification and quantification of anti-drug antibodies
ORR | up to 24 month
  Overall response rate assessed by the investigator according to RECIST version 1.1
DCR | up to 24 month
  Disease control rate assessed by the investigator according to RECIST version 1.1
PFS | up to 24 month
  Progression-free survival assessed by the investigator according to RECIST version 1.1
TTR | up to 24 month
  Time to response assessed by the investigator according to RECIST version 1.1
DOR | up to 24 month
  Duration of response assessed by the investigator according to RECIST version 1.1

CONTACTS AND LOCATIONS:
Locations (2):
- Australia (2):
  - Macquarie University Hospital, North Ryde, New South Wales
  - Cabrini Malvern Hospital, Malvern, Victoria